CLINICAL TRIAL: NCT00968695
Title: Clinical Trial on the Effects of Long Term Administration of 20% Albumin in the Cardiovascular and Renal Function, And Hepatic Hemodynamics in Advanced Patients With Cirrhosis and Ascites.
Brief Title: Effects of Long Term Albumin 20% Administration in Patients With Cirrhosis and Ascites.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Organization: Grifols Therapeutics LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IG0802
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Cirrhosis; Ascites
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Albumin (Experimental): The subjects will be receiving albumin 20% infusions
  Interventions: Drug: Albumin

INTERVENTIONS:
Drug: Albumin — The pattern of administration of 20% human albumin is 1.5g/kg every week to be infused in 6 hours with a minimum of 90g up and a maximum of 150g in patients weighing less than 60 kg and more than 100 kg, respectively. Treatment duration is 12 weeks, which are 13 administrations of albumin.
  Other Names: Albutein 20%

SUMMARY:
Effects of long term albumin administration on the cardiocirculatory and renal function and hepatic hemodynamics in patients with advanced cirrhosis and ascites.

DETAILED DESCRIPTION:
Pharmacodynamic study of pathophysiological nature to assess the effects of prolonged administration of human albumin in the cardiocirculatory and renal function and hepatic hemodynamics in patients with advanced cirrhosis and ascites.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years and less than 80 years.
* Diagnosis of liver cirrhosis by biopsy or by clinical, laboratory, or ultrasound.
* Daily requirement of diuretics at least 200mg of spironolactone or 100mg of spironolactone and 40 mg of furosemide
* Renal dysfunction defined by a plasma concentration of serum creatinine ≥ 1.2 mg / dl, blood urea nitrogen ≥ 25 mg / dl or a serum sodium concentration ≤ 130 mEq / L.

Exclusion Criteria:

* Refractory Ascites (paracentesis requirements over 1 month.
* Neoplastic disease including liver cancer if it exceeds the Milan criteria (one nodule> 5 cm or three nodules> 3 cm).
* History of transjugular intrahepatic portosystemic shunt (TIPS) or surgical shunt
* Gastrointestinal bleeding or bacterial infection documented in the past 15 days.
* Heart failure or structural heart disease.
* Organic renal insufficiency(proteinuria, hematuria and / or ultrasound data nephropathy).
* Moderate or severe lung chronic disease.
* Transplant.
* Infection with human immunodeficiency virus.
* Active addiction to drugs.
* Mental state that prevents the patient understand the nature, extent and consequences of the study, except for hepatic encephalopathy.
* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To asses change from Baseline plasma renin concentration at Week 14 | 14 weeks
  Plasma renin activity will be measured at Baseline and Week 14
To asses change from Baseline plasma renin concentration at Week 20 | 20 weeks
  Plasma renin activity will be measured at Baseline and Week 20
To asses change from Baseline plasma concentration of noradrenaline at week 14 | 14 weeks
  Plasma noradrenaline concentration will be measured at Baseline and Week 14
To asses change from Baseline plasma concentration of noradrenaline at Week 20 | 20 weeks
  Plasma noradrenaline concentration will be measured at Baseline and Week 20
To assess change from Baseline glomerular filtration rate at Week 14 | 14 weeks
  Glomerular filtration rate will be measured at Baseline and Week 14
To assess change from Baseline glomerular filtration rate at Week 20 | 20 weeks
  Glomerular filtration rate will be measured at Baseline and Week 20
To assess change from Baseline cardiac output at Week 14 | 14 weeks
  Cardiac output will be measured at Baseline and Week 14
To assess change from Baseline cardiopulmonary pressures at Week 14 | 14 weeks
  Cardiopulmonary pressures will be measured at Baseline and Week 14
To assess change from Baseline free hepatic pressure at Week 14 | 14 weeks
  Free hepatic pressure will be measured at Baseline and Week 14
To assess change from Baseline wedged hepatic pressure at Week 14 | 14 weeks
  Wedged hepatic pressure will be measured at Baseline and Week 14
To assess change from Baseline echocardiography at Week 14 | 14 weeks
  Echocardiography will be measured at Baseline and Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Arroyo, MD, Principal Investigator — Hospital Clínic of Barcelona
Locations (6):
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clínic of Barcelona, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez J, Claria J, Amoros A, Aguilar F, Castro M, Casulleras M, Acevedo J, Duran-Guell M, Nunez L, Costa M, Torres M, Horrillo R, Ruiz-Del-Arbol L, Villanueva C, Prado V, Arteaga M, Trebicka J, Angeli P, Merli M, Alessandria C, Aagaard NK, Soriano G, Durand F, Gerbes A, Gustot T, Welzel TM, Salerno F, Banares R, Vargas V, Albillos A, Silva A, Morales-Ruiz M, Carlos Garcia-Pagan J, Pavesi M, Jalan R, Bernardi M, Moreau R, Paez A, Arroyo V. Effects of Albumin Treatment on Systemic and Portal Hemodynamics and Systemic Inflammation in Patients With Decompensated Cirrhosis. Gastroenterology. 2019 Jul;157(1):149-162. doi: 10.1053/j.gastro.2019.03.021. Epub 2019 Mar 22. PMID 30905652